CLINICAL TRIAL: NCT04472819
Title: A Phase I, Randomized, Double -Blinded, Placebo-Controlled, Single and Multiple Dose and Food Effect Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of SHR2285 Tablets in Healthy Subjects
Brief Title: The Single, Multiple Dose and Food Effect Study of SHR2285 Tablets on Pharmacokinetics and Pharmacodynamics in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR2285-104
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SHR2285 Part 1A (Experimental): Participant received one of 7 dose levels of SHR2285 tablet as single-dose oral administration
  Interventions: Drug: SHR2285 tablet
- Placebo Part 1A (Placebo Comparator): Single ascending doses of placebo orally
  Interventions: Drug: Placebo
- SHR2285 Part 1B (Experimental): Participant received one dose of SHR2285 tablet as single-dose oral administration
  Interventions: Drug: SHR2285 tablet
- Placebo Part 1B (Placebo Comparator): Single doses of placebo orally
  Interventions: Drug: Placebo
- SHR2285 Part 2 (Experimental): Participant received one of 4 dose levels of SHR2285 tablet as multi-dose oral administration
  Interventions: Drug: SHR2285 tablet
- Placebo Part 2 (Placebo Comparator): Multiple ascending doses of placebo orally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR2285 tablet — single dose or multi-dose
  Arms: SHR2285 Part 1A; SHR2285 Part 1B; SHR2285 Part 2
Drug: Placebo — single dose or multi-dose
  Arms: Placebo Part 1A; Placebo Part 1B; Placebo Part 2

SUMMARY:
The study is a randomized, doubled-blinded, placebo-controlled, Phase I trials. The study is divided into two parts. The first part is a single-dose escalated study (SAD,part 1A ) and food effect study (SAD, part 1B ) in healthy subjects. The second part is a multi-dose escalated study (MAD) in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects, aged 18-55 (including boundary);
2. Body mass index (BMI) between 18 to 28 kg/m2 (including boundary), male body weight ≥50 kg and <90 kg , female body weight ≥45kg and <90kg;
3. Participant with no clinically significant findings in vital signs, physical examination, 12-lead ECG ,X-ray and laboratory parameters.
4. Understand the study procedures and methods, voluntary to participate in the study and signed the informed consent.

Exclusion Criteria:

1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) or total bilirubin/direct bilirubin > upper limit of normal (ULN) during screening/baseline.
2. Serum creatinine> ULN during screening/baseline.
3. Positive faecal occult blood
4. Abnormal coagulation function.
5. A clinical history of coagulation dysfunction; subjects with adverse reaction of antiplatelet drugs or anticoagulant drugs.
6. Subjects with severe head trauma or head surgery within 2 years or surgery within 3 months prior to the screening.
7. Blood donation or blood loss within 1 month≥200 mLor≥400 mL within 3 months before administration.
8. Human immunodeficiency virus antibody, syphilis serological examination, hepatitis b virus surface antigen, hepatitis c virus antibody were positive.

9.3 months prior to screening involved in any drug or medical device clinical studies or within 5 half-life of drugs before screening.

10.Female subjects who did not receive contraception at least 30 days before administration and etc.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and severity of adverse events. | Part 1: Pre-dose to day 7 after single dose administration and Part 2: Pre-dose to day 14after multiple dose administration
Maximum observed serum concentration (Cmax) for Food Effect of SHR2285 on pharmacokinetics parameters in healthy subjects. | Part 1A: Pre-dose to day 7 after single dose administration and Part 1B: Pre-dose to day 7 after single dose administration
Time to maximum observed serum concentration (Tmax) for Food Effect of SHR2285 on pharmacokinetics parameters in healthy subjects. | Part 1A: Pre-dose to day 7 after single dose administration and Part 1B: Pre-dose to day 7 after single dose administration
Time to elimination half-life (T1/2) for Food Effect of SHR2285 on pharmacokinetics parameters in healthy subjects. | Part 1A: Pre-dose to day 7 after single dose administration and Part 1B: Pre-dose to day 7 after single dose administration
Area under the plasma concentration versus time curve (AUC0-last) for Food Effect of SHR2285 on pharmacokinetics parameters in healthy subjects. | Part 1A: Pre-dose to day 7 after single dose administration and Part 1B: Pre-dose to day 7 after single dose administration

SECONDARY OUTCOMES:
Maximum observed serum concentration (Cmax) for single dose of SHR2285. | Part 1:Pre-dose to day 3 after single dose administration and Part 2:Pre-dose to day 9 after multiple dose administration
Time to maximum observed serum concentration (Tmax) for single dose of SHR2285. | Part 1:Pre-dose to day 3 after single dose administration and Part 2:Pre-dose to day 9 after multiple dose administration
Time to elimination half-life (T1/2) for single dose of SHR2285. | Part 1:Pre-dose to day 3 after single dose administration and Part 2:Pre-dose to day 9 after multiple dose administration
Area under the plasma concentration versus time curve (AUC0-last) for single dose of SHR2285. | Part 1:Pre-dose to day 3 after single dose administration and Part 2:Pre-dose to day 9 after multiple dose administration
Steady-state peak concentration (Cmax，ss) for multiple dose of SHR2285. | Pre-dose to day 9 after multiple dose administration
Steady state valley concentration (Ctrough，ss) for multiple dose of SHR2285. | Pre-dose to day 9 after multiple dose administration.
Accumulation ratio (Racc) for multiple dose of SHR2285. | Pre-dose to day 9 after multiple dose administration
Clotting factor XI (FXI) activity . | Part 1:Pre-dose to day 7 after single dose administration and Part 2:Pre-dose to day 14 after multiple dose administration
Change of activated partial thromboplastin time (APTT) from baseline. | Part 1:Pre-dose to day 7 after single dose administration and Part 2:Pre-dose to day 14 after multiple dose administration
Change of prothrombin time (PT) from baseline. | Part 1:Pre-dose to day 7 after single dose administration and Part 2:Pre-dose to day 14 after multiple dose administration
Change of international normalization ratio (INR) from baseline. | Part 1:Pre-dose to day 7 after single dose administration and Part 2:Pre-dose to day 14 after multiple dose administration

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu J, Zhao N, Huang J, Li J, Zhao X, Xiang Q, Yang S, Dong Y, Wang H, Li Y, Yang G, Cui Y. The Safety, Pharmacokinetics, and Pharmacodynamics of SHR2285, an Oral Small Molecule Factor XIa Inhibitor, in Healthy Chinese Volunteers. Clin Drug Investig. 2023 Jun;43(6):435-445. doi: 10.1007/s40261-023-01281-8. Epub 2023 Jun 16. PMID 37326942